CLINICAL TRIAL: NCT06132386
Title: Analysis of Cellular Kinases and Aging in PBMCs and Colorectal Tissue
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00307426; R56AI161030-01A1 (NIH); R01AG064908-03 (NIH)
Record Dates: First submitted 2023-10-20; First posted 2023-11-15 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections; Aging
Keywords: tenofovir; pharmacokinetic; cellular kinase
MeSH Terms: conditions — HIV Infections | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — rectal tissue and blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers, not taking Tenofovir (TFV) based PrEP
  Interventions: Other: biopsy
- Healthy volunteers, steady state Tenofovir (TFV) based regimen
  Interventions: Other: biopsy
- Persons infected with HIV taking Tenofovir (TFV) and emtricitabine (FTC) based HIV treatment
  Interventions: Other: biopsy

INTERVENTIONS:
Other: biopsy — colorectal biopsy for tissue acquisition

SUMMARY:
The goal of this clinical study is to learn about the effect of aging on certain enzymes, or proteins, in the blood and colon. The study involves collection of blood and colon tissue biopsies using a flexible sigmoidoscope or colonoscope. This study is also investigating how medications tenofovir and emtricitabine interact with certain enzymes. The investigators will compare the difference in enzyme activity between people taking tenofovir and emtricitabine, to those who are not taking tenofovir and emtricitabine.

DETAILED DESCRIPTION:
This project involves obtaining peripheral blood mononuclear cells (PBMCs) and colorectal tissue samples from study participants in order to measure adenylate kinase 2 (AK2) and muscle-type creatine kinase (CKM) enzyme levels in various age populations. Both AK2 and CKM has been demonstrated to be vital enzymes in converting the prodrug tenofovir (TFV) into its active form, tenofovir diphosphate (TFV-DP). However, no study has yet investigated the effect of aging on AK2 or CKM in tissues relevant to HIV infection and prevention. This study will investigate the AK2 and CKM variability in individuals from various age groups and how the pharmacokinetics (PK) of tenofovir (TFV) vary with altering levels of cellular enzymes in different age populations

ELIGIBILITY:
Inclusion Criteria:

1. English speaking male or female volunteers between the ages of 18-50 for younger adults or 65-80 for older adults
2. Willing to provide written informed consent
3. Willing to abstain from insertion of anything in rectum for 72 hours before and 72 hours after the endoscopic procedure for colorectal tissue collection.
4. Not currently participating in other research studies involving drugs and/or medical devices.

For participants not infected with HIV (Control Cohort A)

1. No known risk for HIV exposure or a documented negative HIV-1/HIV-2 Ag/Ab test in the past 3 months (HIV risk, but not on PrEP)
2. Documented negative HBsAg in those taking study TFV (i.e. cohort B)

For participants not infected with HIV, but taking or willing to take TFV (PrEP Cohort B)

1. Currently taking TFV-based oral PrEP daily or willing to take oral TFV-containing PrEP for one week
2. Documented negative HIV-1/HIV-2 Ag/Ab test in the past 3 months
3. Documented negative HBsAg

For participants infected with HIV (ARV Cohort C)

1. Virologically suppressed HIV for at least 6 months prior to screening.
2. Taking tenofovir disoproxil fumarate or tenofovir alafenamide containing regimen to treat HIV

Exclusion Criteria:

1. History of inflammatory bowel disease or active inflammatory condition of the GI tract
2. History of significant gastrointestinal bleeding
3. Current medically-indicated use of warfarin or heparin or other anticoagulant medications associated with increased risk for bleeding following mucosal biopsy (e.g., daily high dose aspirin [>81 mg], non-steroidal anti-inflammatory drugs [NSAIDs], or Pradaxa®)
4. Use of systemic immunomodulatory medications within 4 weeks of enrollment
5. Use of rectally administered medications within 4 weeks of enrollment
6. Use of product containing nonoxynol-9 within 4 weeks of enrollment
7. Use of any investigational products within 4 weeks of enrollment
8. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease.
9. Active rectal infection (GC, Chlamydia, HSV). Participants screening positive for GC/CT at the time of endoscopy will be excluded from analysis (and replaced).

   For participants not undergoing a concurrent endoscopic procedure for indication unrelated to this study:
10. Hct <36%
11. Platelet count <150/mm3
12. International normalised ratio blood test > 1.2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population include adults between the ages of 18-50 and 65-80. The population recruited will include healthy volunteers and persons on HIV treatment or prevention that contains tenofovir.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three cohorts of participants will be recruited, with younger adults (18-50 years old) and older adults (65-80 years old) in each cohort.
Groups:
- HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (18-50 Years); HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (18-50 Yrs); HIV Negative, Steady State Tenofovir (TFV) Based Regimen (18-50 Years); HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (65-80 Years); HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65-80 Yrs); HIV Negative, Steady State Tenofovir (TFV) Based Regimen (65-80 Years): biopsy: colorectal biopsy for tissue acquisition
Period: Overall Study
Arm/Group | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (18-50 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (18-50 Yrs) | HIV Negative, Steady State Tenofovir (TFV) Based Regimen (18-50 Years) | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (65-80 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65-80 Yrs) | HIV Negative, Steady State Tenofovir (TFV) Based Regimen (65-80 Years)
Started | 11 | 1 | 0 | 3 | 6 | 0
Completed | 10 | 0 | 0 | 3 | 5 | 0
Not Completed | 1 | 1 | 0 | 0 | 1 | 0
Not completed — ineligble laboratory | 1 | 0 | 0 | 0 | 1 | 0
Not completed — ineligible vital signs | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No healthy volunteers on Steady-state Tenofovir were enrolled.
Groups:
- HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (18 - 50 Years); HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (18 - 50 Yrs); HIV Negative, Steady State Tenofovir (TFV) Based Regimen (18 - 50 Years); HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (65 - 80 Years); HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65 - 80 Yrs); HIV Negative, Steady State Tenofovir (TFV) Based Regimen (65 - 80 Years): biopsy: colorectal biopsy for tissue acquisition
- Total: Total of all reporting groups
Arm/Group | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (18 - 50 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (18 - 50 Yrs) | HIV Negative, Steady State Tenofovir (TFV) Based Regimen (18 - 50 Years) | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (65 - 80 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65 - 80 Yrs) | HIV Negative, Steady State Tenofovir (TFV) Based Regimen (65 - 80 Years) | Total
Number analyzed (Participants) | 11 | 1 | 0 | 3 | 6 | 0 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 1 | 0 | 0 | 0 | 0 | 12
  >=65 years | 0 | 0 | 0 | 3 | 6 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 0 | 2 | 0 | 0 | 7
  Male | 7 | 0 | 0 | 1 | 6 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0 | 0 |  | 0
  Asian | 1 | 0 |  | 0 | 0 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0 | 0 |  | 0
  Black or African American | 1 | 1 |  | 1 | 2 |  | 5
  White | 9 | 0 |  | 2 | 4 |  | 15
  More than one race | 0 | 0 |  | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0 | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 1 |  | 3 | 6 |  | 21

OUTCOME MEASURES:

1. Primary Outcome: Concentration of AK2 in Colorectal Tissue
Description: Concentration in nanometers (nm) of AK2 in colorectal tissue.
Time Frame: Once within one month
Population: Only participants who completed the rectal tissue biopsy are included in the analysis population.
Measure: Median (Inter-Quartile Range); unit: nm
Groups:
- HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FC) Based HIV Treatment (18-50 Years); HIV Negative, Steady State Tenofovir (TFV) Based Regimen (18-50 Years); HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (65-80 Years); HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65-80 Yrs); HIV Negative, Steady State Tenofovir (TFV) Based Regimen (65-80 Years): biopsy: colorectal biopsy for tissue acquisition
Arm/Group | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (18-50 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FC) Based HIV Treatment (18-50 Years) | HIV Negative, Steady State Tenofovir (TFV) Based Regimen (18-50 Years) | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (65-80 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65-80 Yrs) | HIV Negative, Steady State Tenofovir (TFV) Based Regimen (65-80 Years)
Number analyzed (Participants) | 10 | 0 | 0 | 3 | 5 | 0
nm | 12232 [11658 to 12951] |  |  | 12975 [11874 to 13731] | 13173 [11767 to 13521] |

2. Primary Outcome: Concentration of CKM in Colorectal Tissue
Description: Concentration in nanometers (nm) of CKM in colorectal tissue
Time Frame: Once within one month
Population: Only participants who completed the rectal tissue biopsy are included in the analysis population.
Measure: Median (Inter-Quartile Range); unit: nm
Groups:
- HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65-80Yrs); HIV Negative, Steady State Tenofovir (TFV) Based Regimen (65-80 Years): biopsy: colorectal biopsy for tissue acquisition
Arm/Group | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (18-50 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (18-50 Yrs) | HIV Negative, Steady State Tenofovir (TFV) Based Regimen (18-50 Years) | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (65-80 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65-80Yrs) | HIV Negative, Steady State Tenofovir (TFV) Based Regimen (65-80 Years)
Number analyzed (Participants) | 10 | 0 | 0 | 3 | 5 | 0
nm | 4143 [3873 to 4554] |  |  | 3236 [3157 to 3920] | 4176 [3750 to 4587] |

3. Primary Outcome: Concentration of AK2 in Peripheral Blood Mononuclear Cells
Description: Concentration in nanometers (nm) of AK2 in peripheral blood mononuclear cells
Time Frame: Once within one month
Population: Only participants who completed the rectal tissue biopsy are included in the analysis population.
Measure: Median (Inter-Quartile Range); unit: nm
Arm/Group | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (18-50 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (18-50 Yrs) | HIV Negative, Steady State Tenofovir (TFV) Based Regimen (18-50 Years) | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (65-80 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65-80 Yrs) | HIV Negative, Steady State Tenofovir (TFV) Based Regimen (65-80 Years)
Number analyzed (Participants) | 10 | 0 | 0 | 3 | 5 | 0
nm | 2035 [1561 to 2458] |  |  | 1175 [558 to 1799] | 1740 [1180 to 2253] |

ADVERSE EVENTS:
Time Frame: From enrollment up to one month
Description: No participants were enrolled in the Healthy Volunteers, steady state Tenofovir (TDF) based regimen, therefore the number of participants at risk for adverse events is zero.
Groups:
- HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (65-80 Years; HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65-80 Yrs): biopsy: colorectal biopsy for tissue acquisition
Arm/Group | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (18-50 Years) | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (18-50 Yrs) | HIV Negative, Not Taking Tenofovir (TFV) Based PrEP (65-80 Years | HIV Positive Taking Tenofovir (TFV) and Emtricitabine (FTC) Based HIV Treatment (65-80 Yrs)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/1 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/1 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/11 | 0/1 | 0/3 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT06132386/Prot_SAP_000.pdf